CLINICAL TRIAL: NCT06435897
Title: Management of Autoimmune Conditions With Mesenchymal Stem Cells (MSCs) and CAR-T Cells
Brief Title: Autoimmune Disease Treatment With Mesenchymal Stem Cells (MSCs) and CAR-T Cells
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-24003
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Autoimmune Diseases
Keywords: CAR-T; MSC; autoimmune disease; autoantibody; B cell; plasma cell; CD19; BCMA
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC combined with 4SCAR T-cell therapy for autoimmune diseases (Experimental): nfusion of 4SCAR T cells at 10^6 cells/kg body weight and MSCs at 3x10^6 cells via IV
  Interventions: Biological: fetal MSCs combined with 4SCAR T cells

INTERVENTIONS:
Biological: fetal MSCs combined with 4SCAR T cells — Infusion of 4SCAR T cells at 10^6 cells/kg body weight and MSCs at 3x10^6 cells via IV

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of mesenchymal stem cells (MSCs) in combination with CAR-T cells in treating autoimmune disease. Another goal of the study is to learn more about the safety and function of the MSCs combined with CAR-T cells and their long term effects in autoimmune disease patients.

DETAILED DESCRIPTION:
Autoimmune disease refers to the disease in which the immune system reacts to the host's own body and causes damage to tissues and organs. At present, the pathogenesis of various autoimmune diseases is still not well understood, but an imbalanced immune tolerance plays a key role in this process.

An ideal therapy to autoimmune disease should eradicate pathogenic autoimmune cells but retain the protective immunity. The chimeric antigen receptor-modified T (CAR-T) cell technology has proven to be highly effective in targeting B cell malignancies, and the treatment-induced B cell and antibody deficiencies have implications for treating autoantibody-related autoimmune diseases. Studies have shown that CAR-T cells targeting B cell surface molecules can kill autoreactive B lymphocytes in pemphigus vulgaris (PV) and systemic lupus erythematosus (SLE) patients. Thus, CAR-T targeting antibody-producing cells has potential in treating autoimmune diseases including PV, SLE, autoimmune hemolytic anemia, Sjogren's syndrome etc..

MSCs have immune modulatory and immunosuppressive effects. MSCs have been extensively studied and clinically evaluated for the treatment of autoimmune diseases and graft versus host disease (GVHD) caused by hematopoietic stem cell transplantation (HSCT). In many studies, MSCs have demonstrated promising beneficial effects that can reduce severe autoimmune reactions. In recent years, MSCs have been used in synergy with CAR-T cells to address the shortcomings of CAR-T cells. Fetal tissue-derived clonal MSCs (fMSCs) have extended expansion potential and express rich levels of various growth factors. The fMSCs also resove a main limitation in MSC quality and reliability issues related to product consistency of MSCs. As such, innovative strategies to maximise the synergistic effects of CAR-Ts and MSCs have been proposed by either using MSCs as a supplementary intervention to assist in CAR-T based immunotherapies or as part of a sequential therapy regimen.

CD19- and BCMA-specific CAR is based on activation of intracellular signalijng domains of T cells by the extracellular single chain variable fragment (scFv) antibodies against CD19 and BCMA. The activated CAR-T cells can target and kill B cells. The investigation plans to use genetically modified T cells to express 4th generation lentiviral CARs with an inducible caspase 9 self-withdrawal gene (4SCAR) to increase the safety of this specific approach. Besides targeting CD19 and BCMA, other B cell and plasma cell surface molecules will also be targeted and included in the treatment design. Based on accumulated experiences, the 4SCAR T cells have shown high safety profile without serious cytokine release syndrome (CRS) or neural toxicities in patients. Through this trial, the safety and long-term efficacy of synergistic B-cell- and plasma-cell-specific 4SCAR T-cell therapy with MSCs will be evaluated, providing clinical evidence to support the use of 4SCAR-T cells and MSCs in the treatment of autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

1. older than 18 years of age.
2. established autoimmune conditions.
3. the KPS score over 80 points, and survival time is more than 3 months.
4. greater than Hgb 80 g/L.
5. no contraindications to blood cell collection.

Exclusion Criteria:

1. accompanied with other active diseases and difficult to assess treatment response.
2. bacterial, fungal, or viral infection, unable to control.
3. living with HIV.
4. active HBV or HCV infection.
5. pregnant and nursing mothers.
6. under systemic steroid treatment within a week of the treatment.
7. prior failed CAR-T treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 1 month
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
Safety of 4SCAR T cells in patients with autoimmune diseases using CTCAE 5 standard to evaluate the level of adverse events | 12 week
  Safety of 4SCAR T cells in patients with autoimmune diseases using CTCAE 5 standard to evaluate the level of adverse events with measuring cytokine response

SECONDARY OUTCOMES:
Number of participants with reduced symptoms or stabilized conditions after treatment assessed by short term clinical effects | 6 months
  Number of participants with reduced symptoms or stabilized conditions after treatment assessed by short term clinical effects using study assessment table.
The activity of 4SCAR T cells in patients with autoimmune diseases | 1 year
  B cell and immunoglobulin suppression activity of 4SCAR T cells in patients with autoimmune diseases
The activity of 4SCAR T cells in patients with autoimmune diseases | 1 year
  CAR copies in patients with autoimmune diseases
The activity of 4SCAR T cells in patients with autoimmune diseases | 1 year year
  The immunoglobulin levels in patients with autoimmune diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No